CLINICAL TRIAL: NCT00793572
Title: Tandem Autologous HCT/Nonmyeloablative Allogeneic HCT From HLA-Matched Related and Unrelated Donors Followed by Bortezomib Maintenance Therapy for Patients With High-Risk Multiple Myeloma
Brief Title: Autologous or Syngeneic Stem Cell Transplant Followed by Donor Stem Cell Transplant and Bortezomib in Treating Patients With Newly Diagnosed High-Risk, Relapsed, or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marco Mielcarek, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2070.00; NCI-2009-01473 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MPI X05251; 2070.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclosporine; Cyclosporins; fludarabine phosphate; Melphalan; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy (Experimental): See Detailed Description
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Bortezomib; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Syngeneic Bone Marrow Transplantation; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo transplantation
  Other Names: Autologous Stem Cell Transplantation
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Cyclosporine — Given IV
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo transplantation
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo transplantation
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Procedure: Syngeneic Bone Marrow Transplantation — Undergo transplantation
Radiation: Total-Body Irradiation — Undergo radiotherapy
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies the side-effects and anti-cancer effects of giving an autologous or syngeneic stem cell transplant followed by an allogeneic donor stem cell transplant and bortezomib. Patients treated on this trial have newly diagnosed high-risk, relapsed, or refractory multiple myeloma (MM). Giving chemotherapy before an autologous stem cell transplant slows or stops the growth of cancer cells by preventing them from dividing or killing them. Stem cells that were harvested earlier from the patient's blood and frozen are then returned to the patient to replace the blood-forming cells that were destroyed by chemotherapy. Giving chemotherapy and total-body irradiation before an allogeneic donor stem cell transplant also prevents the patient's immune system from rejecting the donor's stem cells. Undergoing an autologous or syngeneic stem cell transplantation followed by an allogeneic donor stem cell transplant and bortezomib may be overall more effective in killing cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Progression-free survival (PFS) at 2 years after the autograft (=< 50% in historic controls).

SECONDARY OBJECTIVES:

I. Overall survival (OS) at 2 years after the autograft.

II. Non-relapse mortality (NRM) at 200 days and 1 year after allograft.

III. Incidence of grades II-IV acute graft-versus-host-disease (GVHD) and chronic extensive GVHD.

IV. Safety of bortezomib maintenance therapy after stem cell transplantation.

OUTLINE:

PERIPHERAL BLOOD STEM CELL (PBSC) MOBILIZATION: Patients undergo PBSC mobilization and collection using the preferred regimens at the participating institution.

CONDITIONING CHEMOTHERAPY AND AUTOLOGOUS OR SYNGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION (HSCT): Patients receive high-dose melphalan intravenously (IV) on day -2 followed by an autologous or syngeneic HSCT on day 0.

NON-MYELOABLATIVE ALLOGENEIC HSCT: Beginning 40-180 days after autologous HSCT, patients receive 1 of the following regimens:

1. HLA-IDENTICAL RELATED DONOR: Patients receive cyclosporine IV or orally (PO) twice daily (BID) starting on days -3 to 56, and taper until day 180. Patients then undergo total-body irradiation (TBI) and non-myeloablative allogeneic HSCT on day 0. Four to six hours after completion of allogeneic HSCT, patients receive mycophenolate mofetil (MMF) PO BID on days 0-27.
2. HLA-UNRELATED DONOR: Patients receive fludarabine phosphate IV on days -4 to -2. Patients also receive cyclosporine IV or PO BID starting on days -3 to 100 and taper until day 180. Patients then undergo TBI and non-myeloablative allogeneic HSCT on day 0. Four to six hours after completion of allogeneic HSCT, patients receive MMF PO thrice daily (TID) on days 0-27 and then BID on days 27-40 with taper of MMF on days 40-96.

MAINTENANCE THERAPY: Beginning 60-120 days after allogeneic HSCT, patients receive bortezomib subcutaneously (SC) on days 1 and 4 of 14-day cycles for 9 months or for up to 18 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients must have received induction therapy (e.g., vincristine, doxorubicin, dexamethasone [VAD], thalidomide/dexamethasone) for a minimum of 4 cycles
* Must have the capacity to give informed consent
* Must have an human leukocyte antigen (HLA) genotypically identical sibling or a phenotypically matched relative or, at a minimum, a high likelihood of identifying an HLA-matched unrelated donor; the determination of availability of a suitable unrelated donor may be based on a World-Book search
* In addition, patients must meet at least one of the criteria A-I (A-G at time of diagnosis or pre-autograft):

  * A) Any abnormal karyotype by metaphase analysis except for isolated t(11,14) and constitutional cytogenetic abnormality
  * B) Fluorescence in situ hybridization (FISH) translocation 4;14
  * C) FISH translocation 14;16
  * D) FISH deletion 17p
  * E) Beta2-microglobulin > 5.5 mg/L
  * F) Cytogenetic hypodiploidy
  * G) Plasmablastic morphology (>= 2%)
* DONOR: HLA genotypically identical sibling or phenotypically matched relative OR
* DONOR: HLA phenotypically matched unrelated donor (according to Standard Practice HLA matching criteria, Grade #2.1)

  * Matched HLA-A, B, C, DRB1, and DQB1 alleles by high resolution typing.
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing

Exclusion Criteria:

* Recurrent or non-responsive (less than partial response [PR]) MM after at least two different lines of conventional chemotherapy
* Progressive MM after a previous autograft
* Life expectancy severely limited by disease other than malignancy
* Seropositive for the human immunodeficiency virus (HIV)
* Females who are pregnant or breastfeeding
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Patients with active non-hematological malignancies (except non-melanoma skin cancers) or those with non-hematological malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within 5 years; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Patients with fungal infection and radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Patients with the following organ dysfunction:

  * Symptomatic coronary artery disease or ejection fraction < 40% or other cardiac failure requiring therapy; myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  * Ejection fraction is required if the patient has a history of anthracyclines or history of cardiac disease
  * Diffusing lung capacity for carbon monoxide (DLCO) < 50%, forced expiratory volume in 1 second (FEV) < 50% and/or receiving supplementary continuous oxygen; the Fred Hutchinson Cancer Research Center (FHCRC) principle investigator (PI) of the study must approve of enrollment of all patients with pulmonary nodules
  * Liver function abnormalities: Patient with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; the patient will be excluded if he/she is found to have fulminant liver failure; cirrhosis of the liver with evidence of portal hypertension; alcoholic hepatitis; esophageal varices; a history of bleeding esophageal varices; hepatic encephalopathy; uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time ascites related to portal hypertension; bacterial or fungal liver abscess; biliary obstruction; chronic viral hepatitis with total serum bilirubin > 3 mg/dL; and symptomatic biliary disease;
  * Karnofsky score < 70% for adult patients
* Patient with poorly controlled hypertension and on multiple antihypertensives
* Patients with current >= grade 2 peripheral neuropathy
* Patient has an active bacterial or fungal infection unresponsive to medical therapy
* DONOR: Identical twin
* DONOR: Donors unwilling to donate PBSC
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness
* DONOR: Failure to meet FHCRC criteria for stem cell donation
* DONOR: Age < 12 years
* DONOR: A positive anti-donor cytotoxic crossmatch
* DONOR: Patient and donor pairs must not be homozygous at mismatched allele

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mielcarek, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241
- [Derived] Green DJ, Maloney DG, Storer BE, Sandmaier BM, Holmberg LA, Becker PS, Fang M, Martin PJ, Georges GE, Bouvier ME, Storb R, Mielcarek M. Tandem autologous/allogeneic hematopoietic cell transplantation with bortezomib maintenance therapy for high-risk myeloma. Blood Adv. 2017 Nov 9;1(24):2247-2256. doi: 10.1182/bloodadvances.2017010686. eCollection 2017 Nov 14. PMID 29296873

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 49.2 [32.8 to 69.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Surviving Progression-free
Description: Number of subjects surviving without progressive disease post-transplant.
  Progressive disease criteria:
  1. Greater than 25% increase in serum (absolute increase must be ≥0.5 g/dL) or urine (absolute increase must be ≥200 mg/24h) M proteins compared to best response status after autologous transplant.
  2. Appearance of new lytic bone lesions or plasmacytomas.
Time Frame: At 2 years after the autograft
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Number analyzed (Participants) | 32
Participants | 14

2. Secondary Outcome: Number of Patients With Grade II-IV Acute GVHD
Description: Number of patients who developed acute GVHD post allogeneic transplant.
  aGVHD Stages
  Skin:
  1. - a maculopapular eruption involving < 25% BSA
  2. - a maculopapular eruption involving 25 - 50% BSA
  3. - generalized erythroderma
  4. - generalized erythroderma w/ bullous formation and often w/ desquamation
  Liver:
  1. - bilirubin 2.0 - 3.0 mg/100 mL
  2. - bilirubin 3 - 5.9 mg/100 mL
  3. - bilirubin 6 - 14.9 mg/100 mL
  4. - bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 2 skin w/ no gut/liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 w/ extreme constitutional symptoms or death
Time Frame: 100 days post allo transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Number analyzed (Participants) | 32
Participants | 14

3. Secondary Outcome: Number of Patients With Chronic GVHD
Description: Number of subjects with classic chronic or chronic extensive GVHD post allogeneic transplant.
Time Frame: 1 year post allo
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Number analyzed (Participants) | 32
Participants | 10

4. Secondary Outcome: Number of Patients With Toxicities Related to Bortezomib Maintenance Therapy
Description: Number of subjects with toxicities related to bortezomib maintenance therapy post-transplant.
Time Frame: Up to 100 days after the autograft or allograft
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Number analyzed (Participants) | 32
Participants | 1

5. Secondary Outcome: Number of Patients With Non-relapse Mortality
Description: Number of subjects with non-relapse mortalities post allogeneic transplant.
Time Frame: 200 and 365 days after allo
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Number analyzed (Participants) | 32
Participants
  200 days post allo | 1
  1 Year post allo | 1

6. Secondary Outcome: Number of Patients Surviving Overall
Description: Number of subjects surviving two years post autologous transplant.
Time Frame: At 2 years after the autograft
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Number analyzed (Participants) | 32
Participants | 21

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100 post Auto; SAEs: Conditioning through Day 200 post Auto
Arm/Group | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy
Serious Adverse Events (participants affected / at risk) | 16/32
Other Adverse Events (participants affected / at risk) | 13/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy (N=32)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Bronchial infection (Infections and infestations) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
GVHD (Immune system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Blood and lymphatic system disorders, Other (Microangiopathy) (Blood and lymphatic system disorders) | 1 (1)
Infections and infestations, Other (Serum) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandem Auto-/Nonmyeloablative Allo-HCT and Maintenance Therapy (N=32)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (5)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes